CLINICAL TRIAL: NCT03773991
Title: Multimodal Assessment of Dyspnea, Cardiopulmonary Structure and Function in Chronic Hemodialysis Patients
Brief Title: Dyspnea Assessment in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Paediatrics, University of Western Ontario. Director of The Lilibeth Caberto Kidney Clinical Research Unit, London Health Sciences Centre., London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 110256
Record Dates: First submitted 2018-11-29; First posted 2018-12-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Dyspnea; Uremic; End Stage Renal Disease; Chronic Lung Disease; Chronic Heart Disease; Hemodialysis-Induced Symptom; Sodium Excess
Keywords: Dyspnea; Hemodialysis; End Stage Renal Disease
MeSH Terms: conditions — Dyspnea; Kidney Failure, Chronic; Hypernatremia | interventions — Echocardiography; Fractional Exhaled Nitric Oxide Testing; Respiratory Function Tests; Blood Specimen Collection; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance Hemodialysis Patients: Patients on chronic hemodialysis therapy due to end-stage renal disease.
  * Proton Lung MRI
  * Sodium MRI of the leg
  * Chest CT
  * Transthoracic Echocardiography
  * Fractional Exhaled Nitric Oxide
  * Six-Minute Walk Test
  * Pulmonary Function Tests
  * Blood sampling
  * Self-administered dyspnea questionnaires
  Interventions: Diagnostic Test: Lung MRI; Diagnostic Test: Sodium MRI; Diagnostic Test: Chest CT; Diagnostic Test: Echocardiography; Diagnostic Test: Fractional Exhaled Nitric Oxide; Diagnostic Test: Pulmonary Function Tests; Diagnostic Test: Blood Sampling; Diagnostic Test: Six-Minute Walk Test; Diagnostic Test: Dyspnea Questionnaires

INTERVENTIONS:
Diagnostic Test: Lung MRI — Proton Lung Magnetic Resonance Imaging
Diagnostic Test: Sodium MRI — Sodium Soft Tissue Magnetic Resonance Imaging
Diagnostic Test: Chest CT — High-resolution Quantitative Chest CT
Diagnostic Test: Echocardiography — Transthoracic 2D Speckle-Tracking Echocardiography
Diagnostic Test: Fractional Exhaled Nitric Oxide — Fractional Exhaled Nitric Oxide testing
Diagnostic Test: Pulmonary Function Tests — Spirometry and Plethysmography
Diagnostic Test: Blood Sampling — Blood testing for: standard-of-care, inflammatory biomarkers, uremic toxins
Diagnostic Test: Six-Minute Walk Test — Six-Minute Walk Test
Diagnostic Test: Dyspnea Questionnaires — Modified Medical Research Council; University of California, San Diego Shortness of Breath Questionnaire; Borg Scale

SUMMARY:
Shortness of breath is very common among patients on dialysis for kidney failure; however, its causes are often not understood. This study will explore the lungs and the heart of these patients to determine the causes of shortness of breath. The amount of salt in the body tissues, which tends to accumulate in dialysis patients and can also cause shortness of breath, will also be measured. Machines that exploit magnetic resonance, ultrasound and x-rays to take images of the body interior will be employed; in addition, breathing tests, questionnaires and blood tests will also be used. 20 patients on dialysis will be recruited and have two visits: one at the beginning of the study and one year later to observe any changes in the lungs, heart and salt accumulation over time.

DETAILED DESCRIPTION:
Rationale:

The available evidence suggest that End-Stage Renal Disease (ESRD) and hemodialysis (HD) have harmful effects on the lungs; the investigators hypothesize that these recurring pulmonary insults, in an analogous way as recurring myocardial ischemic injury for the heart, cause long term impairment in the pulmonary parenchyma, airways and circulation. In addition, observational studies have reported that dyspnea is a common symptom among ESRD patients on chronic HD treatment; however, no study up to now has directly addressed the issue, so that the relationship between dyspnea and pulmonary involvement in the HD population remains poorly understood.

The aim of this study is to explore the pathophysiological basis of dyspnea in patients with end stage renal disease on chronic HD, by using state-of-the-art imaging and functional study techniques.

Study Design:

This is an exploratory study involving a single center recruiting patients from the prevalent dialysis population of London, Ontario. 20 patients on maintenance hemodialysis will be recruited. The patients will undergo imaging, functional studies and blood sampling at the Robarts Research Institute on a non-dialysis day, during the short interval in the dialysis schedule, at baseline and after one year.

Study Procedures:

Blood Collection: blood will be collected from a venous access for standard-of-care tests, uremia and inflammation biomarkers.

Dyspnea Assessment: dyspnea will be assessed with the following self-administered questionnaires: Modified Medical Research Council Breathlessness Scale, the University of California, San Diego Shortness of Breath Questionnaire Pulmonary Function Tests: spirometry and plethysmography pre and post salbutamol administration, carbon monoxide diffusion (DLCO) and the fractional exhaled nitric oxide (FeNO) will be evaluated.

Six Minute Walk Test: the subjects able to do so will perform a six minute walk test, their dyspnea and overall fatigue at baseline and at the end of the exercise will be evaluated using the Borg Scale.

Lung MRI: a proton MRI with ultrashort echo time (UTE) acquisition sequences for the study of lung parenchyma and lung water will be employed. Images will be acquired twice, both pre and post a bronchodilator (salbutamol) challenge.

Sodium MRI: a proton T1 weighted fast-low-angle-shot (FLASH)- sequence will be acquired to delineate the anatomy of the lower leg. Then, a sodium MRI study of the subjects' legs (~5 cm below the knee) will be obtained with the custom-made sodium coil at 3.0 Tesla.

Water content will also be quantified using proton-MRI with fat-suppressed inversion recovery sequence with proton density contrast.

Chest CT: a high-resolution chest CT scan will be performed using a 64-slice CT scanner. A low radiation dose protocol will be employed. A qualitative and quantitative evaluation of pulmonary airways, blood vessels and parenchyma will be performed.

2D Transthoracic Echocardiography: images will be taken in the left lateral decubitus. Images and loops from standard parasternal long axis and short axis, subcostal, apical 4, 2 and 3- chamber views will be recorded and analyzed for: global longitudinal strain, left ventricular ejection fraction, left ventricular mass, left atrial volume, right ventricular diameter, right atrial volume, right ventricular wall thickness, tricuspid annular plane systolic excursion, pulmonary artery systolic pressure, E/A ratio, E/E' ratio at the basal interventricular septum, aortic, mitral, tricuspid and pulmonary valve qualitative and quantitative function.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years.
* Dialysis vintage equal to or greater than 3 months.

Exclusion Criteria

* Smoking history of more than 10 packs/year.
* Active tobacco and/or cannabis smoking.
* Diagnosed chronic pulmonary disease.
* Severe heart failure (NYHA class IV)
* Active infection (including tuberculosis) or malignancy.
* Pregnancy.
* Inability to give consent or understand written information.
* Peripheral oxygen saturation (by pulse oxymetry) dropping below 80% when performing a 12-seconds breathhold.
* Inability to perform spirometry or plethysmography maneuvers.
* Inability to tolerate MRI due to patient size and/or known history of claustrophobia.
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients for this trial will be recruited from incident and prevalent hemodialysis patients receiving care for their kidney disease from the Dialysis Service at London Health Sciences Centre, London Ontario. Up to 20 eligible patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Baseline Modified Medical Research Council scale score. | Baseline
  Baseline dyspnea measured by Modified Medical Research Council scale. 0-4 from lowest (no dyspnea) to highest (most severe dyspnea).
Baseline University of California, San Diego Shortness of Breath Questionnaire score. | Baseline
  Baseline dyspnea measured by University of California, San Diego Shortness of Breath Questionnaire.
  0-120 from lowest (no dyspnea) to highest (most severe dyspnea).
Baseline pulmonary artery diameter. | Baseline
  Baseline pulmonary artery diameter (in millimeters) by chest Computed Tomography.
Baseline lung total blood vessel volume. | Baseline
  Baseline lung total blood vessel volume in ml by chest Computed Tomography.
Baseline lung total airway count. | Baseline
  Baseline lung total airway count by chest Computed Tomography.
Baseline lung low attenuation area. | Baseline
  Baseline lung low attenuation area by chest Computed Tomography.
Baseline lung water content. | Baseline
  Baseline lung water content in arbitrary units measured by proton Magnetic Resonance Imaging.
Baseline soft tissue sodium content. | Baseline
  Baseline soft tissue sodium content in mmol/L measured by sodium Magnetic Resonance Imaging.

SECONDARY OUTCOMES:
One year changes in Modified Medical Research Council scale score. | Baseline and one year
  Comparison of dyspnea measured by Modified Medical Research Council scale at one year versus baseline.
  0-4 from lowest (no dyspnea) to highest (most severe dyspnea).
Correlation between baseline modified Medical Research Council scale score and one year morbidity. | Baseline and one year
  One year morbidity risk by modified Medical Research Council scale baseline score.
Correlation between baseline modified Medical Research Council scale score and one year mortality. | Baseline and one year
  One year mortality risk by modified Medical Research Council scale baseline score.
Correlation between modified Medical Research Council scale score and soft tissue sodium content. | Baseline and one year
  Correlation coefficient between soft tissue sodium content (mmol/L) and modified Medical Research Council scale score.
Correlation between modified Medical Research Council scale score and pulmonary artery diameter. | Baseline and one year
  Correlation coefficient between modified Medical Research Council scale score and pulmonary artery diameter (in millimeters), measured by chest Computed Tomography.
Correlation between modified Medical Research Council scale score and lung total blood vessel volume. | Baseline and one year
  Correlation coefficient between modified Medical Research Council scale score and lung total blood vessel volume (in milliliters), measured by chest Computed Tomography.
Correlation between modified Medical Research Council scale score and lung total airway count. | Baseline and one year
  Correlation coefficient between modified Medical Research Council scale score and lung total airway count, measured by chest Computed Tomography.
Correlation between modified Medical Research Council scale score and lung low attenuation areas. | Baseline and one year
  Correlation coefficient between modified Medical Research Council scale score and lung low attenuation areas, measured by chest Computed Tomography.
Correlation between modified Medical Research Council scale score and lung total water content. | Baseline and one year
  Correlation coefficient between modified Medical Research Council scale score and lung total water content (in arbitrary units), measured by proton Magnetic Resonance Imaging.
One year changes in University of California, San Diego Shortness of Breath Questionnaire score. | Baseline and one year
  Comparison of dyspnea measured by University of California, San Diego Shortness of Breath Questionnaire at one year versus baseline.
  0-120 from lowest (no dyspnea) to highest (most severe dyspnea).
Correlation between baseline University of California, San Diego Shortness of Breath Questionnaire score and one year morbidity. | Baseline and one year
  One year morbidity risk by University of California, San Diego Shortness of Breath Questionnaire baseline score.
Correlation between baseline University of California, San Diego Shortness of Breath Questionnaire score and one year mortality. | Baseline and one year
  One year mortality risk by University of California, San Diego Shortness of Breath Questionnaire baseline score.
Correlation between University of California, San Diego Shortness of Breath Questionnaire score and pulmonary artery diameter. | Baseline and one year
  Correlation coefficient between University of California, San Diego Shortness of Breath Questionnaire score and pulmonary artery diameter (in millimeters), measured by chest Computed Tomography.
Correlation between University of California, San Diego Shortness of Breath Questionnaire score and soft tissue sodium content. | Baseline and one year
  Correlation coefficient between soft tissue sodium content (mmol/L) and University of California, San Diego Shortness of Breath Questionnaire score.
Correlation between University of California, San Diego Shortness of Breath Questionnaire score and lung total blood vessel volume. | Baseline and one year
  Correlation coefficient between University of California, San Diego Shortness of Breath Questionnaire score and lung total blood vessel volume (in milliliters), measured by chest Computed Tomography.
Correlation between University of California, San Diego Shortness of Breath Questionnaire score and lung total airway count. | Baseline and one year
  Correlation coefficient between University of California, San Diego Shortness of Breath Questionnaire score and lung total airway count, measured by chest Computed Tomography.
Correlation between University of California, San Diego Shortness of Breath Questionnaire score and lung low attenuation areas. | Baseline and one year
  Correlation coefficient between University of California, San Diego Shortness of Breath Questionnaire score and lung low attenuation areas, measured by chest Computed Tomography.
Correlation between University of California, San Diego Shortness of Breath Questionnaire score and lung total water content. | Baseline and one year
  Correlation coefficient between University of California, San Diego Shortness of Breath Questionnaire score and lung total water content (in arbitrary units), measured by proton Magnetic Resonance Imaging.
One year changes in lung total blood vessel volume. | Baseline and one year
  Comparison of lung total blood vessel volume (in milliliters) at one year versus baseline, measured by chest Computed Tomography.
One year changes in lung total airway count. | Baseline and one year
  Comparison of lung total airway count at one year versus baseline, measured by chest Computed Tomography.
One year changes in lung water content. | Baseline and one year
  Comparison of lung water content (in arbitrary units) at one year versus baseline, measured by proton Magnetic Resonance Imaging.
One year changes in lung low attenuation areas. | Baseline and one year
  Comparison of lung low attenuation areas at one year versus baseline, measured by chest Computed Tomography.
One year changes in pulmonary artery diameter. | Baseline and one year
  Comparison of pulmonary artery diameter (in millimeters) at one year versus baseline, measured by chest Computed Tomography.
Baseline pulmonary artery systolic pressure. | Baseline
  Baseline pulmonary artery systolic pressure (in mmHg), measured by transthoracic doppler echocardiography.
One year changes in pulmonary artery systolic pressure. | Baseline and one year
  Comparison of pulmonary artery systolic pressure in mmHg at one year versus baseline, measured by transthoracic doppler echocardiography.
Baseline fractional exhaled nitric oxide. | Baseline
  Baseline fractional exhaled nitric oxide measured (in parts per billion).
One year changes in fractional exhaled nitric oxide. | Baseline and one year
  Comparison of fractional exhaled nitric oxide measured (in parts per billion) at one year versus baseline.
Baseline forced expiratory volume at one second/forced vital capacity ratio. | Baseline
  Baseline forced expiratory volume at one second/forced vital capacity ratio by pulmonary function tests.
One year changes in forced expiratory volume at one second/forced vital capacity ratio. | Baseline and one year
  Comparison of forced expiratory volume at one second/forced vital capacity ratio at one year versus baseline, by pulmonary function tests.
Baseline diffusing capacity of the lung for carbon monoxide. | Baseline
  Baseline diffusing capacity of the lung for carbon monoxide (in ml/min/kPa), by pulmonary function tests.
One year changes in diffusing capacity of the lung for carbon monoxide. | Baseline and one year
  Comparison of diffusing capacity of the lung for carbon monoxide (in ml/min/kPa) at one year versus baseline, by pulmonary function tests
Baseline six minute walk distance. | Baseline
  Baseline six minute walk distance (in meters) measured by six minute walk test.
One year changes in six minute walk distance. | Baseline and one year
  Comparison of six minute walk distance (in meters) at one year versus baseline, measured by six minute walk test.
One year changes in soft tissue sodium content. | Baseline and one year
  Comparison of soft tissue sodium content (in mmol/L) at one year versus baseline, measured by sodium Magnetic Resonance Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murtagh FE, Addington-Hall JM, Edmonds PM, Donohoe P, Carey I, Jenkins K, Higginson IJ. Symptoms in advanced renal disease: a cross-sectional survey of symptom prevalence in stage 5 chronic kidney disease managed without dialysis. J Palliat Med. 2007 Dec;10(6):1266-76. doi: 10.1089/jpm.2007.0017. PMID 18095805
- [Background] Fairshter RD, Vaziri ND, Mirahmadi MK. Lung pathology in chronic hemodialysis patients. Int J Artif Organs. 1982 Mar;5(2):97-100. PMID 7095887
- [Background] Zoccali C, Torino C, Tripepi R, Tripepi G, D'Arrigo G, Postorino M, Gargani L, Sicari R, Picano E, Mallamaci F; Lung US in CKD Working Group. Pulmonary congestion predicts cardiac events and mortality in ESRD. J Am Soc Nephrol. 2013 Mar;24(4):639-46. doi: 10.1681/ASN.2012100990. Epub 2013 Feb 28. PMID 23449536
- [Background] Nascimento MM, Qureshi AR, Stenvinkel P, Pecoits-Filho R, Heimburger O, Cederholm T, Lindholm B, Barany P. Malnutrition and inflammation are associated with impaired pulmonary function in patients with chronic kidney disease. Nephrol Dial Transplant. 2004 Jul;19(7):1823-8. doi: 10.1093/ndt/gfh190. Epub 2004 May 18. PMID 15150347
- [Background] Wallin CJ, Jacobson SH, Leksell LG. Subclinical pulmonary oedema and intermittent haemodialysis. Nephrol Dial Transplant. 1996 Nov;11(11):2269-75. doi: 10.1093/oxfordjournals.ndt.a027147. PMID 8941589
- [Background] Bolignano D, Rastelli S, Agarwal R, Fliser D, Massy Z, Ortiz A, Wiecek A, Martinez-Castelao A, Covic A, Goldsmith D, Suleymanlar G, Lindholm B, Parati G, Sicari R, Gargani L, Mallamaci F, London G, Zoccali C. Pulmonary hypertension in CKD. Am J Kidney Dis. 2013 Apr;61(4):612-22. doi: 10.1053/j.ajkd.2012.07.029. Epub 2012 Nov 17. PMID 23164943
- [Background] Barak M, Nakhoul F, Katz Y. Pathophysiology and clinical implications of microbubbles during hemodialysis. Semin Dial. 2008 May-Jun;21(3):232-8. doi: 10.1111/j.1525-139X.2008.00424.x. Epub 2008 Mar 18. PMID 18363602
- [Background] Plesner LL, Warming PE, Nielsen TL, Dalsgaard M, Schou M, Host U, Rydahl C, Brandi L, Kober L, Vestbo J, Iversen K. Chronic obstructive pulmonary disease in patients with end-stage kidney disease on hemodialysis. Hemodial Int. 2016 Jan;20(1):68-77. doi: 10.1111/hdi.12342. Epub 2015 Aug 5. PMID 26245152
- [Background] Pabst S, Hammerstingl C, Hundt F, Gerhardt T, Grohe C, Nickenig G, Woitas R, Skowasch D. Pulmonary hypertension in patients with chronic kidney disease on dialysis and without dialysis: results of the PEPPER-study. PLoS One. 2012;7(4):e35310. doi: 10.1371/journal.pone.0035310. Epub 2012 Apr 18. PMID 22530005
- [Background] Herrero JA, Alvarez-Sala JL, Coronel F, Moratilla C, Gamez C, Sanchez-Alarcos JM, Barrientos A. Pulmonary diffusing capacity in chronic dialysis patients. Respir Med. 2002 Jul;96(7):487-92. doi: 10.1053/rmed.2002.1346. PMID 12194631
- [Background] Kovacevic P, Stanetic M, Rajkovaca Z, Meyer FJ, Vukoja M. Changes in spirometry over time in uremic patients receiving long-term hemodialysis therapy. Pneumologia. 2011 Jan-Mar;60(1):36-9. PMID 21545062
- [Background] McIntyre CW, Odudu A. Hemodialysis-associated cardiomyopathy: a newly defined disease entity. Semin Dial. 2014 Mar;27(2):87-97. doi: 10.1111/sdi.12197. PMID 24738144
- [Background] Belem LC, Zanetti G, Souza AS Jr, Hochhegger B, Guimaraes MD, Nobre LF, Rodrigues RS, Marchiori E. Metastatic pulmonary calcification: state-of-the-art review focused on imaging findings. Respir Med. 2014 May;108(5):668-76. doi: 10.1016/j.rmed.2014.01.012. Epub 2014 Feb 6. PMID 24529738
- [Background] Incalzi RA, Corsonello A, Pedone C, Battaglia S, Paglino G, Bellia V; Extrapulmonary Consequences of COPD in the Elderly Study Investigators. Chronic renal failure: a neglected comorbidity of COPD. Chest. 2010 Apr;137(4):831-7. doi: 10.1378/chest.09-1710. Epub 2009 Nov 10. PMID 19903974
- [Background] Romoff MS, Keusch G, Campese VM, Wang MS, Friedler RM, Weidmann P, Massry SG. Effect of sodium intake on plasma catecholamines in normal subjects. J Clin Endocrinol Metab. 1979 Jan;48(1):26-31. doi: 10.1210/jcem-48-1-26. No abstract available. PMID 422701